CLINICAL TRIAL: NCT04006808
Title: A Reactogenicity, Safety and Immunogenicity Study of GSK's Paediatric Herpes Zoster Subunit Candidate Vaccine (PED-HZ/su) GSK143713A in Immunocompromised Paediatric Renal Transplant Recipients
Brief Title: A Study to Test GlaxoSmithKline's (GSK) Candidate Vaccine-GSK1437173A for Prevention of Shingles in Children With Kidney Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 200075; 2019-000607-33 (EudraCT Number)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PED-HZ/su 12-17 Group (Experimental): Paediatric renal transplant recipients aged 12 to 17 years old, receiving 2 doses of the investigational vaccine (PED HZ/su)
  Interventions: Biological: PED-HZ/su
- Control 12-17 Group (No Intervention): Paediatric renal transplant recipients aged 12 to 17 years old, not receiving the investigational vaccine but being treated according to the local standard of care
- PED-HZ/su 1-11 Group (Experimental): Paediatric renal transplant recipients aged 1 to 11 years old, receiving 2 doses of the investigational vaccine (PED HZ/su).
  Enrolment into this group will be in a staggered manner. Following enrolment into the PED-HZ/su 12-17 group, a safety evaluation of data collected up to visit month 2 will be performed. Upon favourable outcome of the evaluation, enrolment into this group will begin.
  Interventions: Biological: PED-HZ/su
- Control 1-11 Group (No Intervention): Paediatric renal transplant recipients aged 1 to 11 years old, not receiving the investigational vaccine but being treated according to the local standard of care

INTERVENTIONS:
Biological: PED-HZ/su — GSK's candidate vaccine- PED-HZ/su. is administered intramuscularly in the deltoid of the non-dominant arm, on a two-dose schedule in the two investigational groups.
  Arms: PED-HZ/su 1-11 Group; PED-HZ/su 12-17 Group

SUMMARY:
The purpose of this study is to evaluate the reactogenicity, safety and immunogenicity of 2 doses of PED-HZ/su, GSK's vaccine candidate for the prevention of Herpes Zoster (HZ) in immunocompromised paediatric renal transplant recipients aged 1-17 years

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s) who, in the opinion of the investigator, can and will comply, with the requirements of the protocol
* Written or witnessed/thumb printed informed consent obtained from the parent(s)/LAR(s) of the subject prior to performance of any study specific procedure.
* Written informed assent obtained from the subjects when applicable according to local requirements.
* A male or female between, and including, 1 and 17 years of age at the time of randomisation (Visit Day 1)
* Body weight ≥ 6 kg/13.23 pounds.
* A subject is eligible if they meet at least one of the following criteria:

  * Documented previous VZV vaccination OR
  * Medically verified varicella (with source documentation) OR
  * Seropositive for VZV prior to transplantation.
* Subjects with renal transplant more than six months (180 days) prior randomization (Visit Day 1)
* Subject who has received an ABO compatible allogeneic renal transplant (allograft).
* Subject with stable renal function with stability defined as <20% variability between the last two creatinine measurements or based on investigator opinion after review of multiple creatinine measurements.
* Subject receiving maintenance immunosuppressive therapy for the prevention of allograft rejection for a minimum of one month (30 days) prior to randomization (Visit Day 1).
* Female subjects of childbearing potential may be enrolled in the study, if the subject

  * has practiced adequate contraception for 30 days prior to Visit Day 1 and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

Medical conditions

* Any primary kidney disease with a high incidence of recurrent primary kidney disease within the allograft
* Evidence of recurrent primary kidney disease within the current allograft
* Previous allograft loss secondary to recurrent primary kidney disease
* History of more than one organ transplanted (that is, kidney-liver, simultaneous double kidney or kidney-other organ(s) transplanted).
* Subjects with an episode of acute allograft rejection over the six months (180 days) prior to enrolment
* Panel Reactive Antibodies (PRA) calculated PRA (cPRA) or Calculated Reaction Frequency (cRF) score that is unknown at the time of transplant
* VZV serostatus unknown prior to transplant
* Subjects with advanced chronic kidney disease
* Evidence of significant proteinuria (≥ 200 g/mol creatinine) believed to be of renal origin (an example of non-renal origin is proteinuria from mucus in a reconstructed bladder)
* Subjects without multiple dialysis options in the event acute or chronic dialysis needed.
* History of unstable or progressive neurological disorder.
* Subjects ≤ 5 years of age with a history of one or more simple or complex febrile seizures
* Subjects > 5 years with history of one or more complex febrile seizures
* Occurrence of a varicella or HZ episode by clinical history within the 6 months (180 days) preceding Visit Day 1
* Any autoimmune disease, with the following exceptions which do not constitute an exclusion criterion:

  * IgA nephropathy
  * Rapidly progressive glomerulonephritis
  * Membranous glomerulonephritis
  * Idiopathic Type I membranoproliferative glomerulonephritis
  * Diabetes mellitus (type 1 and 2) with diabetic nephropathy
* Confirmed or suspected Human Immunodeficiency Virus or primary immunodeficiency disease
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
* Any condition which, in the judgement of the investigator would make intramuscular injection unsafe.
* Atypical Haemolytic Uraemic Syndrome.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before Visit Day 1 (Day -29 to Day -1), or planned use during the study period.
* Subject in receipt of treatment for rejection during the six months (180 days) prior to enrolment.
* Use of anti-CD20 or other B-cell monoclonal antibody agents within 1 year of Visit Day 1 or planned administration during the duration of the study.
* Administration of blood products 3 months (90 days) prior to Visit Day 1 or planned administration during the duration of the study.
* Administration of immunoglobulins 6 months (180 days) prior to Visit Day 1 or planned administration of immunoglobulins during the duration of the study.
* Administration or planned administration of a vaccine within 30 days prior to Visit Day 1 up to Visit Month 2 with the exception of an inactivated or subunit influenza vaccine which may be given 8 days prior to or 14 days after Visit Day 1 and 8 days prior to or 14 days after Visit Month 1.
* Previous vaccination against HZ
* Varicella vaccination within the 6 months (180 days) preceding Visit Day 1
* Planned administration during the study of an HZ or varicella vaccine (including an investigational or non-registered vaccine) other than the study vaccine

Prior/Concurrent clinical study experience

• Concurrent or planned participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product

* available locally through compassionate use programs,
* submitted for and pending local/country registration,
* approved and registered for use in other countries with well-documented Summary of Product Characteristics or Prescribing Information
* The name of the active component(s) of these immunosuppressants must be provided in the concomitant medication listing

Other exclusions

* Child in care
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) between one month (30 days) prior to Visit Day 1 through two months (60 days) after Visit Month 1.
* Evidence or high suspicion, in the opinion of the investigator, of non-compliance or non-adherence to use of induction and/or maintenance immunosuppressive therapies.
* Failure to fully complete the 7-day pre-vaccination diary card distributed at the Pre-vaccination visit

  * Completion must cover the 7 days immediately prior to randomisation (Visit Day 1).
  * Completion is defined as a minimum of 6 days completed.
  * Subjects with less than 6 days completed may be offered a new date for Visit Day 1 and the opportunity to comply with the completion of the 7-day pre-vaccination diary card prior to the new planned Visit Day 1.
* Any study personnel or their immediate dependants, family, or household member.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects from the interventional groups, with solicited local adverse events (AEs) | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  Assessed solicited local AEs are pain, redness and swelling at the injection site. Pain includes tenderness.
  Note: GSK diary cards for collecting solicited local and general AEs/symptoms is different for subjects < 6 years and ≥ 6 years. Hence the age category of 1-11 years is further split to 1-5 years and 6-11 years.
Number of subjects from the interventional groups, with solicited general AEs | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  Assessed solicited general AEs among Infants/Toddlers/Children < 6 years are:
  * Drowsiness
  * Fever*
  * Irritability/Fussiness
  * Loss of appetite
  * Gastrointestinal (GI) symptoms**
  Assessed solicited general AEs among Children ≥ 6 years are:
  * Fatigue
  * Fever*
  * GI symptoms**
  * Headache
  * Myalgia
  * Shivering (chills)
    * Fever is defined as temperature ≥ 38.0°C/100.4°F **GI symptoms include nausea, vomiting, diarrhoea, and/or abdominal pain Note: GSK diary cards for collecting solicited local and general AEs/symptoms is different for subjects < 6 years and ≥ 6 years. Hence the age category of 1-11 years is further split to 1-5 years and 6-11 years.
Number of subjects from the control groups with solicited general symptoms | Within 7 days after Visit Day 1
  Assessed solicited general symptoms among Infants/Toddlers/Children < 6 years are:
  * Drowsiness
  * Fever*
  * Irritability/Fussiness
  * Loss of appetite
  * GI symptoms**
  Assessed solicited general symptoms among Children ≥ 6 years are:
  * Fatigue
  * Fever*
  * GI symptoms**
  * Headache
  * Myalgia
  * Shivering (chills)
    * Fever is defined as temperature ≥ 38.0°C/100.4°F **GI symptoms include nausea, vomiting, diarrhoea, and/or abdominal pain As subjects from the control group are not vaccinated, they will not complete the diary card for local solicited symptoms.
Number of subjects from the control groups with solicited general symptoms | Within 7 days after Visit Month 1
  Assessed solicited general symptoms among Infants/Toddlers/Children < 6 years are:
  * Drowsiness
  * Fever*
  * Irritability/Fussiness
  * Loss of appetite
  * GI symptoms**
  Assessed solicited general symptoms among Children ≥ 6 years are:
  * Fatigue
  * Fever*
  * GI symptoms**
  * Headache
  * Myalgia
  * Shivering (chills)
    * Fever is defined as temperature ≥ 38.0°C/100.4°F **GI symptoms include nausea, vomiting, diarrhoea, and/or abdominal pain
Number of subjects from the interventional groups with unsolicited AEs after each vaccination | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects from the control groups with unsolicited symptoms | Within 30 days after Visit Day 1
  An unsolicited symptom is any symptom reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects from the control groups with unsolicited symptoms | Within 30 days after Visit Month 1
  An unsolicited symptom is any symptom reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects with serious adverse events (SAEs), potential immune mediated diseases (pIMDs) and biopsy confirmed renal allograft rejection. | From Visit Day 1 up to Visit Month 2
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity.
  pIMDs are sub sets of Adverse events of special interest (AESIs) that include autoimmune disease and other inflammatory and/neurological disorders of interest, which may or may not have autoimmune aetiology.
  The renal allograft rejections are biopsy confirmed pathophysiological changes indicative of rejection. The rejection is graded for severity and extent of histologic inflammation and injury. The reporting period for any renal allograft rejection is from Visit Day 1 to the study end (month 2).
Number of subjects from the interventional groups with seizures | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  All seizures occurring within 30 days following study vaccination are reported.
Number of subjects from the non-interventional groups with seizures | Within 30 days after Visit Day 1
  All seizures occurring within 30 days after visit day 1 are reported, for the control groups.
Number of subjects from the non-interventional groups with seizures | Within 30 days after Visit Month 1
  All seizures occurring within 30 days of visit month 1 are reported, for the control groups
Number of subjects from the interventional groups with generalized convulsive seizures | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure.
Number of subjects from the non-interventional groups with generalized convulsive seizures | Within 7 days after Visit Day 1
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure
Number of subjects from the non-interventional groups with generalized convulsive seizures | Within 7 days after Visit Month 1
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure
Percentage of subjects with Anti-gE antibody concentrations in terms of Geometric Mean Concentrations (GMCs) | At Month 2 (one-month post-dose 2)
  The geometric mean concentration (GMC) calculations are performed by taking the anti log of the mean of the log concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value equal to half the cut-off for GMC calculation

SECONDARY OUTCOMES:
Number of subjects with SAEs, pIMDs and biopsy confirmed renal allograft rejections from day 1 to month 13 | From Visit Day 1 up to Visit Month 13
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity pIMDs are sub sets of Adverse events of special interest (AESIs) that include autoimmune disease and other inflammatory and/neurological disorders of interest, which may or may not have autoimmune aetiology.
  The renal allograft rejections are biopsy confirmed pathophysiological changes indicative of rejection. The rejection is graded for severity and extent of histologic inflammation and injury.
  This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)
Occurrence of Herpes Zoster cases | From Visit Day 1 until Visit Month 13
  HZ may present classically with a unilateral, dermatomal rash that is associated with pain, pruritus, allodynia or other altered sensation. In this population, disseminated HZ may occur and present with a generalized rash with systemic symptoms such as fever. All children enrolled in the trial have a history of primary VZV infection or vaccination and in the presence of immunosuppression, disseminated HZ cannot be distinguished clinically from varicella This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)
Number of subjects from the interventional pooled age group with solicited local AEs | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years.
  The assessed local AEs solicited are:
  * Pain
  * Redness
  * Swelling Note: Pain includes tenderness.
Number of subjects from the interventional pooled age group with solicited general AEs | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years.
  The assessed solicited general AEs among Infants/Toddlers/Children < 6 years are:
  * Drowsiness
  * Fever*
  * Irritability/Fussiness
  * Loss of appetite
  * Gastrointestinal (GI) symptoms**
  The assessed solicited general AEs among Children ≥ 6 years are:
  * Fatigue
  * Fever*
  * GI symptoms**
  * Headache
  * Myalgia
  * Shivering (chills)
    * Fever is defined as temperature ≥ 38.0°C/100.4°F **GI symptoms include nausea, vomiting, diarrhoea, and/or abdominal pain
Number of subjects from the non-interventional pooled age group with solicited general symptoms | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years.
  The assessed solicited general symptoms among Infants/Toddlers/Children < 6 years are:
  * Drowsiness
  * Fever*
  * Irritability/Fussiness
  * Loss of appetite
  * GI symptoms**
  The assessed solicited general symptoms among Children ≥ 6 years are:
  * Fatigue
  * Fever*
  * GI symptoms**
  * Headache
  * Myalgia
  * Shivering (chills)
    * Fever is defined as temperature ≥ 38.0°C/100.4°F **GI symptoms include nausea, vomiting, diarrhoea, and/or abdominal pain As subjects from the control group are not vaccinated, they will not complete the diary card for local solicited symptoms.
Number of subjects from the interventional pooled age group with unsolicited AEs after each vaccination | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years. An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects from the non-interventional pooled age group with unsolicited symptoms | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years. An unsolicited symptom is any symptom reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects from the non-interventional pooled age group with unsolicited symptoms | Within 30 days after Visit Month 1
  The pooled age group includes all subjects aged 1-17 years. An unsolicited symptom is any symptom reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited adverse event.
Number of subjects from the pooled age groups with any SAEs, pIMDs and biopsy confirmed renal allograft rejections | From Visit Day 1 until Visit Month 2
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity pIMDs are sub sets of Adverse events of special interest (AESIs) that include autoimmune disease and other inflammatory and/neurological disorders of interest, which may or may not have autoimmune aetiology.
  The renal allograft rejections are biopsy confirmed pathophysiological changes indicative of rejection. The rejection is graded for severity and extent of histologic inflammation and injury.
Number of subjects from the pooled age groups with any SAEs, pIMDs and biopsy confirmed renal allograft rejections | From Visit Day 1 until Visit Month 13
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity pIMDs are sub sets of Adverse events of special interest (AESIs) that include autoimmune disease and other inflammatory and/neurological disorders of interest, which may or may not have autoimmune aetiology.
  The renal allograft rejections are biopsy confirmed pathophysiological changes indicative of rejection. The rejection is graded for severity and extent of histologic inflammation and injury.
Number of subjects from the pooled age groups with HZ | From Visit Day 1 until Visit Month 13
  HZ may present classically with a unilateral, dermatomal rash that is associated with pain, pruritus, allodynia or other altered sensation. In this population, disseminated HZ may occur and present with a generalized rash with systemic symptoms such as fever. All children enrolled in the trial have a history of primary VZV infection or vaccination and in the presence of immunosuppression, disseminated HZ cannot be distinguished clinically from varicella.
  This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)
Number of subjects from the interventional pooled age group with seizures | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years. All seizures occurring within 30 days following study vaccination are reported
Number of subjects from the non-interventional pooled age group with seizures | Within 30 days after Visit Day 1
  The pooled age group includes all subjects aged 1-17 years. All seizures occurring with 30 days after visit day 1 are reported
Number of subjects from the non-interventional pooled age group with seizures | Within 30 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years. All seizures occurring with 30 days after visit month 1 are reported
Number of subjects from the interventional pooled age group with generalized convulsive seizures | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years.
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure
Number of subjects from the non-interventional pooled age group with generalized convulsive seizures | Within 7 days after each vaccination (vaccines administered on day 1 and month 1)
  The pooled age group includes all subjects aged 1-17 years.
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure
Number of subjects from the non-interventional pooled age group with generalized convulsive seizures | Within 7 days after Visit Month 1
  The pooled age group includes all subjects aged 1-17 years.
  Generalized convulsive seizures are classified as follows:
  * Level 1 of diagnostic certainty: witnessed sudden loss of consciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 2 of diagnostic certainty: history of unconsciousness AND generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations
  * Level 3 of diagnostic certainty: history of unconsciousness AND other generalized motor manifestations
  * Level 4 of diagnostic certainty: reported generalized convulsive seizure with insufficient evidence to meet the case definitions for Level 1, 2 or 3 of diagnostic certainty above
  * Level 5 of diagnostic certainty: Not a case of generalized convulsive seizure Only levels 1 to 3 of generalized convulsive seizures will comprise the analysis for this outcome measure
Vaccine Response Rate (VRR) for Anti-glycoprotein (Anti-gE) antibody concentrations | At Month 2 and Month 13
  The Vaccine Response Rate for anti-gE antibodies is defined as the percentage of subjects who have at least:
  * a 4-fold increase in the post-dose 2 anti-gE Ab concentration as compared to the pre-vaccination anti-gE Ab concentration, for subjects who are seropositive at baseline, or,
  * a 4-fold increase in the post-dose 2 anti-gE Ab concentration as compared to the anti-gE Ab cut-off value for seropositivity, for subjects who are seronegative at baseline.
  This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)
Median fold increase of anti-gE antibody concentrations | At Month 2 and Month 13
  Median fold increase in antibody concentration with 95% Confidence Interval is tabulated for the interventional groups by age strata (1-11 years and 12-17 years) This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)
Percentage of subjects with anti-gE antibody concentrations in terms of GMCs | At Day 1 (pre-vaccination) and Month 13
  GMC calculations are performed by taking the anti log of the mean of the log concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value equal to half the cut-off for GMC calculation
Percentage of subjects in the interventional pooled age group, with Anti-gE antibody concentrations in terms of GMCs | At Day 1, Month 2 and Month 13
  GMC calculations are performed by taking the anti log of the mean of the log concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value equal to half the cut-off for GMC calculation.
  Median fold increase in antibody concentration with 95% Confidence Interval is to be tabulated for the interventional groups by pooled age category (1-17 years).
  This outcome measure is analysed during epoch 002 (day 1 to month 2) and during epoch 003 (month 2- month 13)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Italy (5):
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Torino
- GSK Investigational Site, Gdansk, Poland
- Spain (5):
  - GSK Investigational Site, BaracaldoVizcaya
  - GSK Investigational Site, Espluges de Llobregat
  - GSK Investigational Site, HebrOn
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- United Kingdom (7):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Glasgow Strathclyde
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Mollo A, Peri M, Lodi L, Gissi A, Lionetti P, Marrani E, Mastrolia MV, Tondo A, Tintori V, Sardi I, Indolfi G, Trapani S, Galli L, Venturini E, Astorino V, Azzari C, Ricci S. Considering recombinant herpes zoster vaccine for fragile pediatric patients: A new opportunity. Vaccine. 2025 Apr 19;53:127072. doi: 10.1016/j.vaccine.2025.127072. Epub 2025 Apr 7. PMID 40198934